CLINICAL TRIAL: NCT05586360
Title: T-reg Function Changes: a Novel Immune Regulatory Effect Underlying Benefit of Statin Use on Lethal Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Michael Marrone, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103472
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Neoadjuvant; Statin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simvastatin (Experimental): Patients randomized to the statin group will receive 40 mg oral simvastatin QD for eight weeks prior to prostatectomy, including the day of surgery.
  Interventions: Drug: Simvastatin 40mg
- Control (No Intervention): Patients randomized to the control group receive no intervention prior to prostatectomy.

INTERVENTIONS:
Drug: Simvastatin 40mg — Simvastatin 40mg taken orally daily for 8 weeks
  Arms: Simvastatin

SUMMARY:
This study will evaluate whether simvastatin reduces intraprostatic immunosuppressive microenvironment through YAP-mediated T-reg dysfunction, and increases intraprostatic anti-tumor immune response in men recently diagnosed with localized prostate cancer electing to receive prostatectomy for their care. Half the men will be randomized to receive statins for 8 weeks prior to their surgery, while the other half will receive standard of care.

DETAILED DESCRIPTION:
Prior research has demonstrated a consistently strong inverse association between statin drug use and risk of developing lethal prostate cancer, and a stronger protective effect with a longer duration of use. Further, in men with clinically localized prostate cancer, statins are associated with a reduced risk of progression to metastasis and dying from prostate cancer. For statins to have clinical utility as chemo-preventive and therapeutic (adjuvant) agents, additional characterization of the mechanisms through which statins interact with the tumor microenvironment are needed. Statin drugs have been shown to inhibit Yes-associated protein (YAP) nuclear translocation and transcriptional activation (via YAP phosphorylation) required for T regulatory cell (T-reg) immunosuppressive function. YAP is a critical regulator of the immunosuppressive microenvironment contributing to T-reg differentiation and immunosuppressive function and antitumor T cell response.

Simvastatin is a moderate intensity statin regimen recommended for cholesterol reduction, and was previously shown to have a strong cytoplasmic YAP sequestration activity. This trial is designed to investigate the effect of 40 mg oral simvastatin daily on YAP-mediate T-reg disfunction and antitumor immune response. Eligible patients include men newly diagnosed with pathologically-confirmed localized prostate cancer determined to be intermediate (stage T2b, or Gleason 7 or PSA 10-20ng/mL) or high risk (stage T2c or PSA >/= 20 ng/mL, or Gleason >/= 8) of biochemical recurrence at the time of biopsy; not currently taking a statin who are scheduled for prostatectomy. For the trial, 52 patients will be randomized in a 1:1 ratio to the statin group or the control group. Randomization sequence will be computer generated using random blocks with concealed allocation of the random treatment assignment (e.g., statin or control) and will be stratified by race (Black vs non-Hispanic White) and BMI (<30 vs ≥30). Patients randomized to the statin group will receive moderate intensity simvastatin (40mg, day) for eight weeks until the date of prostatectomy. Patients randomized to the control group will not receive any intervention, this is not a placebo-controlled trial and participants, and investigators will not be masked. Patients in both groups will receive standard clinical laboratory assessments at baseline and at the end of the study after eight weeks to evaluated adherence based on the change in cholesterol and inflammation biomarkers from baseline to the end of follow-up at eight weeks. Multiplex immunofluorescence will be used to assess intra-prostatic YAP-mediate T-reg dysfunction (the number FOXP3+ T-regs with phosphorylated YAP), and intra-prostatic anti-tumor immune response (the count and density of CD4+ and CD8+ T cells) in whole tumor sections obtained from the tumor block containing the index tumor (i.e., largest and/or highest Gleason sum).

ELIGIBILITY:
Inclusion Criteria:

1. Men with pathologically-confirmed localized prostate cancer determined to be intermediate (stage T2b, or Gleason 7, or PSA 10-20 ng/mL) or high risk (stage T2c, or PSA >/=20 ng/mL, or Gleason >/=8) of biochemical recurrence at the time of biopsy
2. Electing to undergo prostatectomy;
3. Ability to provide written informed consent and willing to complete study procedures.

Exclusion Criteria:

1. Current statin use or use of non-statin lipid-lowering drug (fibrates, bile acid sequestrants, or niacin);
2. Current use of medications contraindicated for concomitant use with 40mg simvastatin:

   * Gemfibrozil
   * Cyclosporine
   * Danazol
   * CYP3A4 inhibitors: itraconazole; ketoconazole; posaconazole; erythromycin; clarithromycin; telithromycin; HIV protease inhibitors; boceprevir; telaprevir; nefazodone
3. Current use of medications requiring lower dose of simvastatin not already listed as exclusions criteria:

   * Verapamil
   * Diltiazem
   * Amiodarone
   * Ranolazine
   * Calcium channel blockers: verapamil; diltiazem; amlodipine
4. Men with low-density lipoprotein cholesterol <50mg/dL
5. Statin use in the previous 12 months;
6. Discontinued statin use because of statin-related adverse event;
7. Evidence or suspicion of metastases;
8. Prior neoadjuvant or adjuvant chemotherapy, hormone therapy, or radiation therapy;
9. History of non-prostate cancer other than non-melanoma skin cancer in the last 24 months;
10. Diagnosed diabetes or currently taking diabetes medications
11. Prior myocardial infarction or stroke
12. Chronic liver disease (hepatitis or cirrhosis) or abnormal liver function (>1.5x clinical laboratory's upper limit of normal alanine aminotransferase);
13. Stage 4 or 5 chronic kidney disease (Creatinine clearance / estimated glomerular filtration rate < 30 mL/min calculated by Cockgroft-Gault formula);
14. History of myopathy or inflammatory muscle disease (>3x clinical laboratory's upper limit of normal creatine kinase).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This trial is focused on prostate cancer, a cancer of a male organ, and is applicable to men only. Men from all racial and ethnic groups are eligible to participate in this trial.
Enrollment: 36 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Intra-prostatic YAP-mediated T-reg dysfunction in total tissue area | 8 weeks
  Number of men diagnosed with localized prostate cancer randomized to receive a statin prior to prostatectomy that have greater intra-prostatic YAP-mediated T-reg dysfunction compared to men randomized to the control group.
  Intra-prostatic T-reg dysfunction will be determined by the proportion of Foxp3+ T-regs with phosphorylated YAP sequestered in the cytoplasm detected by multiplex immunofluorescence and digital quantitative image analysis.

SECONDARY OUTCOMES:
Intra-prostatic YAP-mediated T-reg dysfunction, limited to tumor infiltrating Tregs | 8 weeks
  Number of men randomized to the statin group that have greater YAP-mediated T-reg dysfunction compared to men randomized to the control group restricting to tumor-infiltrating T-regs only.
  Intra-prostatic T-reg dysfunction will be determined by the proportion of Foxp3+ T-regs with phosphorylated YAP sequestered in the cytoplasm detected by multiplex immunofluorescence and digital quantitative image analysis.
Intra-prostatic YAP-mediated T-reg dysfunction, limited to T-regs in adjacent normal and stromal tissue | 8 weeks
  Number of men randomized to the statin group that have greater YAP-mediated T-reg dysfunction compared to men randomized to the control group restricting to the subset of T-regs in the adjacent normal and stromal tissue area.
  Intra-prostatic T-reg dysfunction will be determined by the proportion of Foxp3+ T-regs with phosphorylated YAP sequestered in the cytoplasm detected by multiplex immunofluorescence and digital quantitative image analysis.
Intra-prostatic anti-tumor immune response | 8 weeks
  Density (cell counts per total area evaluated) of CD4,+ CD8+, PD-1+, and CTLA-4+ T cells, and PD-L1+ tumor cells detected by multiplex immunofluorescence and digital quantitative image analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marrone, PhD, Principal Investigator — Public Health Sciences
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina